CLINICAL TRIAL: NCT03409133
Title: Feasibility of Neural Feedback for Lower Limb Amputees
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Collaborators: Case Western Reserve University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ronald Triolo, Senior Research Career Scientist, US Department of Veterans Affairs,, Louis Stokes VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 15046-H27
Record Dates: First submitted 2017-12-15; First posted 2018-01-24 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Amputation
Keywords: prosthesis user; phantom sensation; sensory feedback; prosthesis; amputee; amputation; limb loss; robotic prosthesis; neuroprosthesis; sensory restoration; robotic; electromyography; EMG; sensation; myoelectric
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stimulating nerve electrodes & intramuscular recording electrodes (Experimental): Fifteen subjects with lower limb amputation will have multi-contact stimulating nerve cuff electrodes implanted around the nerves in their residual limb. These electrodes will be connected to temporary percutaneous leads.
  During experimental testing, a small amount of electrical current will be delivered to the nerves through multi-contact nerve cuff electrodes.
  Participants also have the option to have recording electrodes implanted within muscles in their lower limb(s). These muscles are associated with prosthetic movement, and recordings from these muscles will be used to develop a controller for a robotic myoelectric prosthesis.
  Interventions: Device: Stimulating nerve electrodes and intramuscular recording electrodes

INTERVENTIONS:
Device: Stimulating nerve electrodes and intramuscular recording electrodes — See Arm Description

SUMMARY:
The purpose of this study is to evaluate the effectiveness of providing sensation of the missing limb to individuals with lower limb loss, including above and below knee amputees. The approach involves delivering small electrical currents directly to remaining nerves via implanted stimulating electrodes. These small electrical currents cause the nerves to generate signals that are then transferred to your brain similar to how information about the foot and lower limb used to be transferred to your brain prior to the amputation.

Individuals also have the option to have recording electrodes implanted within muscles of the lower limb(s) in an attempt to develop a motor controller that would enable the user to have intuitive control of a robotic prosthetic leg.

DETAILED DESCRIPTION:
Electrodes are surgically implanted on one to four nerves of the residual limb. An external wearable device controls the delivery of electrical pulses to the implanted system. The participant will be asked to verbally describe the perceived sensations and highlight their locations on a drawing of a foot presented to them on an electronic screen. An instrumented prosthesis will be developed such that perceived sensations would correspond to prosthesis interactions with the floor. This instrumented prosthesis, also known as a sensory neuroprosthesis, will be worn while the participant is engaging in various functional tasks, such as standing, walking, or climbing stairs, or with visual or mental distractions.

Intramuscular recording electrodes can be implanted in the lower limb(s) and/or hip muscles in order to obtain electromyography (EMG) signals. The EMG recordings from the residual muscles will be used to develop an algorithm which can operate an advanced robotic prosthesis in which the movement of the joint(s) could be controlled.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or greater
* Chronic, medically stable ( > 3 months) unilateral trans-tibial or trans-femoral amputation at the time of implant surgery.
* Potential user of trans-tibial or trans-femoral prostheses for standing or walking
* Viable target nerves in the lower extremity as determined by standard-of-care clinical tests of nerve conduction, response to stimulation, sensory evoked potentials and the like
* Good skin integrity and personal hygiene
* Absence of autoimmune deficiencies, seizure disorders or cardiac abnormalities contraindicating stimulation
* Sufficient social support and personal ability to tolerate study procedures and comply with follow-up schedule

Exclusion Criteria:

* Uncontrolled diabetes to a degree that would preclude surgery
* Significant vascular disease
* Chronic skin ulcerations
* Significant history of poor wound healing
* Significant history of uncontrolled infections
* Active infection
* Significant pain in the residual or phantom limb
* Pregnancy
* Inability to speak English
* Expectation that MRI will be required at any point for the duration of study or while percutaneous leads are in place
* Severe neurological conditions that significantly impair balance or mobility to an extent that independent ambulation is impossible without assistance ( as determined by a healthcare provider)
* Appropriate body habitus (height and weight within acceptable limits as determined by study physician)
* Poor surgical candidate
* Psychiatric or cognitive conditions that could affect cooperation or understanding of instructions and willingness to undergo psychological evaluation, if recommended by study surgeons or investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-11-05 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Stimulation Thresholds | 9 months post implant
  Quantify the minimum stimulation required to evoke electrically induced sensations on the phantom limb.
Functional Gait Assessment (FGA) | 1 year post implant
  The Functional Gait Assessment is a 10 task test that measures postural stability. Each task is scored from 0 -3 with 0 indicating severe impairment in the task and 3 indicating normal ambulation. The scores are combined to give a total score. The maximum score is 30. A higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Triolo, PhD, Principal Investigator — Louis Stokes VA Medical Center
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in neuroprostheses and amputee research. The shared data will be coded, with no PHI included. Approval of the request by local IRB and review of the PI(s) are prerequisites to the sharing of data with the requesting party.
Supporting Information: SAP, Analytic Code
Time Frame: Upon request, IPD sharing will begin 6 months after publication and will be available for up to 1 year. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of the request. Based on the extent of the request, written approvals from local IRB and execution of a Data Sharing Agreement (DSA) might be prerequisite. For more information or to submit a request, please contact Aarika.Sheehan@va.gov.

REFERENCES:
- [Derived] Sheehan A, Siu R, Schmitt M, Vala J, Wright J, Kim D, Li S, Graczyk E, Triolo RJ, Charkhkar H. Impact of Long-Term Home and Community Use of a Lower Limb Sensory Neuroprosthesis. Res Sq [Preprint]. 2025 Sep 19:rs.3.rs-7412528. doi: 10.21203/rs.3.rs-7412528/v1. PMID 41001531